CLINICAL TRIAL: NCT01013064
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Dose Escalation Study of the Safety, Pharmacodynamics and Pharmacokinetics of Single Intravenous Doses of HM10760A in Healthy Adult Korean Subjects
Brief Title: A Study of HM10760A (Long-acting Erythropoietin (EPO)) in Healthy Korean Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-HM10760A-102
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Erythropoietin; Long acting; EPO

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort1 (Experimental)
  Interventions: Drug: HM10760A or Placebo
- Cohort2 (Experimental)
  Interventions: Drug: HM10760A or Placebo
- Cohort3 (Experimental)
  Interventions: Drug: HM10760A or Placebo
- Cohort4 (Experimental)
  Interventions: Drug: HM10760A or Placebo
- Cohort5 (Experimental)
  Interventions: Drug: HM10760A or Placebo
- Cohort6 (Experimental)
  Interventions: Drug: HM10760A or Placebo

INTERVENTIONS:
Drug: HM10760A or Placebo — 0.04 mcg/kg to 2.0mcg/kg once intravenously

SUMMARY:
Study design:

* Randomized, double-blind, placebo-controlled, sequential dose escalation
* Six ascending dose cohorts are planned

Primary Objective:

* To evaluate the safety profile of single escalating intravenous dose levels of HM10760A

DETAILED DESCRIPTION:
Secondary objectives:

* To evaluate the dose response relationship of a single IV dose of HM10760A on pharmacodynamic parameters including hemoglobin, reticulocyte count, and reticulocyte hemoglobin content
* To evaluate the pharmacokinetic profiles of single IV dose levels of HM10760A
* To determine the pharmacologically active dose(PAD) of HM10760A
* To assess the immunogenicity of a single IV dose of HM10760A

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 55 years
* Able and willing to provided written informed consent
* Hemoglobin < 16 g/dL

Exclusion Criteria:

* Prior exposure to EPO, darbepoetin, other EPO support proteins
* hypersensitivity to EPO, darbepoetin, E.coli derived proteins
* Hemoglobinopathy
* SBP > 140 mmHg or < 90 mmHg or DBP > 95 mmHg
* Chronic, uncontrolled, or symptomatic inflammatory disease
* Malignancy(except non-melanoma skin cancer)

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety data, including physical examinations, laboratory evaluation, ECGs, vital signs, adverse events, and immunogenicity | 84 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Clinical, Seoul, South Korea